CLINICAL TRIAL: NCT02734680
Title: Intraoperative Radiotherapy(IORT) Followed by Concurrent Chemoradiotherapy(CCRT) or Stereotactic Radiotherapy(SBRT) for Locally Advanced Pancreatic Cancer
Brief Title: IORT Followed by CCRT or SBRT for Locally Advanced Pancreatic Cancer
Acronym: IFCSLAPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chengfeng Wang, Director of Department of Abdominal Surgical Oncolgoy, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC2015L11
Record Dates: First submitted 2016-04-07; First posted 2016-04-12 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Intraoperative radiotherapy(IORT); Postoperative radiochemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chemoradiotherapy; Radiosurgery; S 1 (combination)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiotherapy(CCRT) Group (Experimental): Concurrent chemoradiotherapy(CCRT) (Total dose: 46 Gy; Single dose: 2 Gy; Frequency: 23; Gemcitabine(GEM), 300 mg/m2 weekly); Followed by taking S-1 orally (40 mg/m2, bid on Day 1-28, Q42d)
  Interventions: Radiation: Concurrent chemoradiotherapy(CCRT); Drug: S-1
- Stereotactic Radiotherapy(SBRT) Group (Experimental): Stereotactic Radiotherapy(SBRT) (Total dose: 45 Gy; Single dose: 3 Gy; Frequency: 15) Followed by taking S-1 orally (40 mg/m2, bid on Day 1-28, Q42d)
  Interventions: Radiation: Stereotactic Radiotherapy(SBRT); Drug: S-1

INTERVENTIONS:
Radiation: Concurrent chemoradiotherapy(CCRT) — Radiation and take gemcitabine(GEM)
  Other Names: Concurrent chemoradiotherapy
  Arms: Concurrent chemoradiotherapy(CCRT) Group
Radiation: Stereotactic Radiotherapy(SBRT) — Stereotactic Radiotherapy(SBRT) (total dose: 45 Gy; single dose: 3 Gy; Frequency:15)
  Other Names: Stereotactic Radiotherapy
  Arms: Stereotactic Radiotherapy(SBRT) Group
Drug: S-1 — Taking S-1 orally after radiation
  Other Names: S-1 orally

SUMMARY:
The purpose of this study is to find the best model of combination of intraoperative radiotherapy(IORT) and postoperative radiochemotherapy for pancreatic cancer.

DETAILED DESCRIPTION:
The trial is funded by Cancer Foundation of China. The trial is prepared to be registered on the clinicaltrail.gov.

Quality assurance plan: every participant is enrolled or excluded by two practiced investigators. And two investigators participated in all steps of the trail, including the record of the data, and the investigators will compare the data. If the data is consistent, the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the workers of research and financial department of National Cancer Center/ Cancer Hospital, Chinese Academy of Medical Sciences.

Data check: the investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms.

Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information, and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 70 participants to take part in the trail. The investigators can recruit about 35 participants every year according to previous experiences, so the investigators should recruit at least for two years.

Plan for missing data: the investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results.

Statistical analysis plan: Kaplan-Meier method would be used to analyze the difference of survival time between the two groups, and the local control rate of the two groups would be compared by chi square test. Statistical analyses would be performed by using IBM SPSS Statistics(version 20; IBM, Chicago, USA). The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as locally advanced pancreatic cancer.
* Cannot be treated by surgical resection.

Exclusion Criteria:

* Treated by chemotherapy or radiotherapy before.
* With distant organ metastasis.
* Cannot tolerate surgery (Intraoperative radiotherapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Overal survival | 2 years
  OS

SECONDARY OUTCOMES:
Disease-specific survival | 2 years
  DSS
Progression-free survival | 2 years
  PFS
Local control rate | 2 years
  LCR

CONTACTS AND LOCATIONS:
Overall Officials: Chengfeng Wang, B.A., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided